CLINICAL TRIAL: NCT02558426
Title: Molecular Analysis of Estrogen Receptors in Patients With Chronic Venous Disease
Brief Title: Estrogen Receptors and Chronic Venous Disease
Acronym: ERCVD
Status: Completed | Type: Observational
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Assistant Professor of Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2013.31
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Estrogen Excess; Varicose Veins
Keywords: Chronic Venous Disease; Estrogen receptors; GPER
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CVD patients: Patients with CVD at various stages (C2-C6 of CEAP classification of CVD) with varicose veins and eligible to receive Open Venous Surgery.
  Interventions: Procedure: Venous Surgery

INTERVENTIONS:
Procedure: Venous Surgery — Patients with Varicose Veins will undergo to venous surgery procedure. Samples obtained from patients undergoing surgical removal of varicose veins will be collected and immediately preserved at -80°. Briefly, the venous tissueswill be excised, homogenized with a motor-driven homogenizer and total RNA will be isolated using the Trizol reagent (Invitrogen, Milan, Italy), according to the manufacturer's instructions. The expression of ERα, ERβ and GPER will be quantified by real-time PCR using the Step OneTM sequence detection system (Applied Biosystems Inc., Milan, Italy), following the manufacturer's instructions

SUMMARY:
Chronic Venous Disease (CVD) is a very common problem affecting western adult population. To date the pathophysiology of CVD development encloses several theories such as the role of extracellular matrix (ECM) components alterations, the alteration of Matrix Metalloproteinases (MMPs) and other related molecules, the endothelial dysfunction, and several genetic factors but none of these could properly explain its genesis. Estrogen Receptors may be involved in CDV pathogenesis. Endogenous estrogens are important regulators of vascular homeostasis and they act mainly via three different ERs which are expressed in the cardiovascular system: ERα, ERβ, and a G protein-coupled estrogen receptor termed GPER. of this study is to explore the expression of estrogen receptors in vessel wall of varicose veins through the entire clinical spectrum of CVD.

DETAILED DESCRIPTION:
Chronic Venous Disease (CVD) is a very common problem affecting western adult population with a prevalence of < 10%, among individuals younger than 30 years for both sex, and with a prevalence of 57% and 77%, in men and women aged ≥ 70 years respectively, and may be frequently associated with other clinical manifestations.

The spectrum of CVD ranges from varicose veins to leg edema, and serious dermal clinical manifestations consisting of hyperpigmentation, eczema, lipodermatosclerosis, and venous skin ulceration.

To date the pathophysiology of CVD development encloses several theories such as the role of extracellular matrix (ECM) components alterations, the alteration of Matrix Metalloproteinases (MMPs) and other related molecules, the endothelial dysfunction, and several genetic factors but none of these could properly explain its genesis.

A recent study (Serra R et al) showed a higher prevalence of CVD among patients with Breast Cancer (BC) respect to general population, especially in those patients that were positive to estrogen receptor (ER) expression.

The presence of ERs was investigated in the walls of normal and varicose veins by Mashiah A. et al, previously, and they documented that increased concentrations of estrogen receptors were found in varicose vein segments respect to healthy controls and this was particularly evident in females.

Endogenous estrogens are important regulators of vascular homeostasis and they act mainly via three different ERs which are expressed in the cardiovascular system: ERα, ERβ, and a G protein-coupled estrogen receptor termed GPER.

Although ERs are also suspected to be involved in the underlying etiology, the exact molecular mechanism responsible for development of CVD as well as the relationship with the wide range of clinical manifestations of CVD remains to be elucidated and the aim of this study is to explore the expression of estrogen receptors in vessel wall of varicose veins collected from patients with varicose veins through the entire clinical spectrum of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Venous Disease and varicose veins eligible to receive open venous surgery procedure

Exclusion Criteria:

* Concomitant Peripheral Artery Disease
* Previous Venous Thromboembolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Venous Disease and varicose veins eligible to receive open venous surgery procedure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
expression of ERα, ERβ and GPER | At month 9th
  The expression of ERα, ERβ and GPER will be quantified by real-time PCR using the Step OneTM sequence detection system (Applied Biosystems Inc., Milan, Italy), following the manufacturer's instructions

REFERENCES:
- [Background] Serra R, Buffone G, de Franciscis A, Mastrangelo D, Molinari V, Montemurro R, de Franciscis S. A genetic study of chronic venous insufficiency. Ann Vasc Surg. 2012 Jul;26(5):636-42. doi: 10.1016/j.avsg.2011.11.036. PMID 22664280
- [Background] Serra R, Buffone G, Costanzo G, Montemurro R, Perri P, Damiano R, de Franciscis S. Varicocele in younger as risk factor for inguinal hernia and for chronic venous disease in older: preliminary results of a prospective cohort study. Ann Vasc Surg. 2013 Apr;27(3):329-31. doi: 10.1016/j.avsg.2012.03.016. Epub 2012 Sep 19. PMID 22998788
- [Background] Serra R, Buffone G, Costanzo G, Montemurro R, Scarcello E, Stillitano DM, Damiano R, de Franciscis S. Altered metalloproteinase-9 expression as least common denominator between varicocele, inguinal hernia, and chronic venous disorders. Ann Vasc Surg. 2014 Apr;28(3):705-9. doi: 10.1016/j.avsg.2013.07.026. Epub 2013 Oct 31. PMID 24184457
- [Background] Serra R, Gallelli L, Buffone G, Molinari V, Stillitano DM, Palmieri C, de Franciscis S. Doxycycline speeds up healing of chronic venous ulcers. Int Wound J. 2015 Apr;12(2):179-84. doi: 10.1111/iwj.12077. Epub 2013 Apr 5. PMID 23557025
- [Background] de Franciscis S, Serra R. Matrix metalloproteinases and endothelial dysfunction: The search for new prognostic markers and for new therapeutic targets for vascular wall imbalance. Thromb Res. 2015 Jul;136(1):5-6. doi: 10.1016/j.thromres.2015.04.022. Epub 2015 Apr 24. No abstract available. PMID 25940670
- [Background] Serra R, Buffone G, Falcone D, Molinari V, Scaramuzzino M, Gallelli L, de Franciscis S. Chronic venous leg ulcers are associated with high levels of metalloproteinases-9 and neutrophil gelatinase-associated lipocalin. Wound Repair Regen. 2013 May-Jun;21(3):395-401. doi: 10.1111/wrr.12035. Epub 2013 Mar 26. PMID 23531093
- [Background] Serra R, Buffone G, Miglietta AM, Abonante S, Giordano V, Renne M, Lugara M, de Franciscis S. Breast cancer and venous disease: a retrospective cohort study. Ann Vasc Surg. 2013 Aug;27(6):762-6. doi: 10.1016/j.avsg.2012.10.020. Epub 2013 Jul 1. PMID 23809843
- [Background] Mashiah A, Berman V, Thole HH, Rose SS, Pasik S, Schwarz H, Ben-Hur H. Estrogen and progesterone receptors in normal and varicose saphenous veins. Cardiovasc Surg. 1999 Apr;7(3):327-31. doi: 10.1016/s0967-2109(98)00132-x. PMID 10386751
- [Background] Meyer MR, Prossnitz ER, Barton M. The G protein-coupled estrogen receptor GPER/GPR30 as a regulator of cardiovascular function. Vascul Pharmacol. 2011 Jul-Sep;55(1-3):17-25. doi: 10.1016/j.vph.2011.06.003. Epub 2011 Jul 5. PMID 21742056